CLINICAL TRIAL: NCT07191990
Title: Evaluation of Post-operative Pain and Bacterial Load Reduction After Application of Different Final Irrigation Protocols in Single Visit Root Canal Treatment of Mandibular First Molar Teeth With Symptomatic Irreversible Pulpitis
Brief Title: Measure Postoperative Pain and Bacterial Reduction After Different Final Irrigation Protocols.
Acronym: PIRRI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Samar Tarek, principal investigator, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SamarRCT01
Record Dates: First submitted 2025-09-03; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Symptomatic Irreversible Pulpitis (SIP)
Keywords: postoperative pain; bacterial load reduction
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Final irrigation by NaOcl at room temperature (Active Comparator): Final irrigation by NaOcl (2.6%) at room temperature 24 °C for 1 min.
  Interventions: Procedure: Final irrigation by NaOcl at room temperature
- Final irrigation by cryotreated NaOcl. (Active Comparator): Final irrigation by cryotreated NaOcl (2.6%) at 2-4 °C for 1 min
  Interventions: Procedure: Final irrigation by cryotreated NaOcl.
- Final irrigation by preheated NaOcl. (Active Comparator): Final irrigation by preheated 60°C(15) NaOcl (2.6%) for 1 min
  Interventions: Procedure: Final irrigation by preheated NaOcl
- Final irrigation with ultrasonic activation of NaOcl. (Active Comparator): Final irrigation with ultrasonic activation of NaOcl(2.6%) for 1 min
  Interventions: Procedure: Final irrigation with ultrasonic activation of NaOcl

INTERVENTIONS:
Procedure: Final irrigation by cryotreated NaOcl. — Final irrigation by cryotreated NaOcl (2.6%) at 2-4 °C for 1 min
  Other Names: cryotreated
  Arms: Final irrigation by cryotreated NaOcl.
Procedure: Final irrigation by preheated NaOcl — Final irrigation by preheated 60°C(15) NaOcl (2.6%) for 1 min.
  Other Names: preheated
  Arms: Final irrigation by preheated NaOcl.
Procedure: Final irrigation with ultrasonic activation of NaOcl — Final irrigation with ultrasonic activation of NaOcl(2.6%) for 1 min
  Arms: Final irrigation with ultrasonic activation of NaOcl.
Procedure: Final irrigation by NaOcl at room temperature — Final irrigation by NaOcl (2.6%) at room temperature 24 °C for 1 min
  Arms: Final irrigation by NaOcl at room temperature

SUMMARY:
The primary objective of root canal treatment is to clean, disinfect, and hermetically seal the root canal system to prevent bacterial penetration; however, postoperative pain is frequently encountered, particularly in patients with symptomatic irreversible pulpitis. This condition, defined by the American Association of Endodontists as an irreversible inflammatory state of the pulp, is commonly associated with spontaneous pain, lingering discomfort, and heightened thermal sensitivity, and often represents a significant challenge in endodontics. Postoperative pain is usually linked to extrusion of microorganisms and debris into the periapical region during chemo-mechanical preparation. Bacteria remain the most persistent pathogens in root canal infections, and although sodium hypochlorite (NaOCl) is considered the most effective irrigant due to its antibacterial and tissue-dissolving properties, complete bacterial elimination before root filling is not always achieved. To enhance its antimicrobial efficacy, various adjunctive approaches have been suggested, including passive ultrasonic activation (PUA) and modifying NaOCl temperature, either by heating or cooling. Cryotherapy has gained increasing attention in endodontics for its potential to decrease postoperative pain and bacterial load, with additional reported benefits in vital pulp therapy, instrumentation, and anesthesia. Previous studies have shown that cryo-irrigation after NaOCl significantly reduces bacterial counts compared to NaOCl alone. Considering the potential benefits of these different irrigation protocols, the present study aims to evaluate and compare their effectiveness in reducing postoperative pain and bacterial load following single-visit root canal treatment of mandibular first molars diagnosed with symptomatic irreversible pulpitis.

The aim of the study will be directed to evaluate postoperative pain and bacterial load reduction after application of different final irrigation protocols in single visit root canal treatment in patients with symptomatic irreversible pulpitis in first molar teeth. this study consists of 60 patients divided into 4 groups each group having 15 patients.

control: Final irrigation by NaOcl (2.6%) at room temperature 24 °C for 1 min interventions: I1: Final irrigation by cryotreated NaOcl (2.6%) at 2-4 °C for 1 min . I2: Final irrigation by preheated 60°C(15) NaOcl (2.6%) for 1 min. I3:Final irrigation with ultrasonic activation of NaOcl(2.6%) for 1 min

ELIGIBILITY:
Inclusion Criteria:

* Patients with age range between 18 to 40.
* No sex predilection.
* Patients with symptomatic irreversible pulpitis.
* Patients able to sign informed consent.
* Restorable teeth
* Positive patient's acceptance for participating in the study.
* Type III distal and mesial canal of first mandibular molar.
* Mild to moderate (5-20) ° curvature according to Schneider

Exclusion Criteria:

* Pregnant females
* Medically compromised patients.
* Patients having analgesics before the treatment
* If antibiotic have been administrated during the past two weeks preoperatively.
* Patients having bruxism or clenching
* Patients having sever malocclusion associated with traumatic occlusion.
* Teeth that have:

Peri-apical periodontitis Root resorption Pain on percussion Pulp stones or calcifications Previous endodontic treatment.

-Non-patent canals

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain after each activation method in comparison to control group | from 6 to 72 hours from the treatment .
  measuring Post-operative pain by Numerical rate scale and pain level will be assigned to one of 4 categorical score: none (0): mild (1-3), severe (7-10).

SECONDARY OUTCOMES:
bacterial load change after final irrigation protocol. | "immediately after the intervention.
  Recording the percentage of bacterial load reduction by collecting samples by paper points, first sample after access cavity and before Root canal treatment.
  second sample after mechanical instrumentation third sample after final irrigation

CONTACTS AND LOCATIONS:
Locations (1):
- Future University in Egypt, Cairo, New Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided